CLINICAL TRIAL: NCT04570956
Title: Phase IIB Randomized Trial of Oral Tamoxifen vs. Topical 4-hydroxytamoxifen Gel vs. Control in Women With Atypical Hyperplasia, Lobular Carcinoma in Situ, or Increased Breast Cancer Risk
Brief Title: Oral Tamoxifen vs. TamGel vs. Control in Women With Atypical Hyperplasia, Lobular Carcinoma In Situ, or Increased Breast Cancer Risk
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: grant and funding expired
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA237607; NCI-2022-02973 (Other: CTRP (Clinical Trials Reporting Program)); 5R01CA237607-05 (NIH); 19-011444 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2020-09-28; First posted 2020-09-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Atypical Hyperplasia; Breast Lobular Carcinoma in Situ; Breast Atypical Lobular Hyperplasia; Breast Carcinoma
MeSH Terms: conditions — Breast Carcinoma In Situ; Breast Neoplasms | interventions — Tamoxifen; Gels

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 2:2:1 with either Oral Tamoxifen 10 mg/day
  * gel placebo, Topical 4-OHT gel 4 mg/each breast/day
  * oral placebo, or Control Oral and gel placebo for 4 weeks of treatment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects with be randomized by MedidataRave and Pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Oral Tamoxifen 10 mg/day (Experimental): Oral Tamoxifen 10 mg/day
  Interventions: Drug: Tamoxifen; Other: Questionnaire Administration
- Topical 4-OHT (4-hydroxytamoxifen) gel 4 mg/each breast/day (Experimental): Topical 4-OHT (4-hydroxytamoxifen) gel 4 mg/each breast/day
  +oral placebo
  Interventions: Drug: Topical 4-OHT( 4-hydroxytamoxifen)gel 4 mg/each breast/day; Other: Questionnaire Administration
- Control (Experimental): Oral and gel placebo
  Interventions: Drug: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Tamoxifen — Oral Tamoxifen 10 mg/day
  Other Names: Oral tamoxifen
  Arms: Oral Tamoxifen 10 mg/day
Drug: Topical 4-OHT( 4-hydroxytamoxifen)gel 4 mg/each breast/day — Topical 4-OHT (4-hydroxytamoxifen) gel 4 mg/each breast/day
  Other Names: Topical gel
  Arms: Topical 4-OHT (4-hydroxytamoxifen) gel 4 mg/each breast/day
Drug: Placebo — placebo pill or placebo gel
  Other Names: placebo pill; placebo gel
  Arms: Control
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
The investigators plan to prospectively study breast tissue changes after a short course of Tamoxifen (Tam).

DETAILED DESCRIPTION:
Women with atypical hyperplasia (AH) and lobular carcinoma in situ (LCIS) are at increased risk of breast cancer (BC) (~1-2 % per year). Over two decades ago, placebo-controlled randomized trials established that oral tamoxifen (20 mg/day) reduces breast cancer risk by 50% in generally defined high risk women, with ~70% reduction in women at high risk specifically due to atypical hyperplasia.[1] Years later, the side effects and toxicity of oral tamoxifen at 20 mg/day remain a significant barrier to its uptake and longterm compliance.[2, 3] To address the issue of toxicity, two main strategies have been pursued: 1) using a lower dose of oral tamoxifen, and 2) using a topical formulation of tamoxifen to avoid systemic side effects. The investigators will perform a prospective study of women with AH or LCIS who will take a short course of prevention therapy; breast tissue samples will be evaluated pre- and post-therapy to identify and evaluate very early biomarkers of response. The overall goal of the study is to evaluate short-term changes in background breast tissue induced by either low-dose oral tamoxifen or topical 4-OHT gel in women with AH or LCIS.

ELIGIBILITY:
Inclusion Criteria:

* Willing to return to enrolling institution for follow-up
* Willing to complete required testing
* Ability to complete questionnaire by themselves or with assistance
* Female (sex that was assigned at birth)
* Ipsilateral intact breast with histology confirmation of atypical ductal or lobular hyperplasia, or lobular carcinoma in situ (LCIS), within the last 12 months, whether surgically excised or not.; OR neither AH nor LCIS but increased breast cancer risk defined as either:

  * Gail model (Breast Cancer Risk Assessment Tool) 5 year breast cancer risk of >= 3%, or
  * International Breast Intervention Study model 10 year breast cancer risk of >= 5%.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%)
* The effects of topical afimoxifene (4-OHT) gel on the developing human fetus at the recommended therapeutic dose are unknown. However, oral tamoxifen is Pregnancy Category D-positive evidence of human fetal risk. For this reason, and because triphenylethylene antiestrogens, including tamoxifen, are known to be teratogenic, women of childbearing potential and their male partners must agree to use at least one effective form of birth control (abstinence is not an allowed method) prior to study entry and for the duration of study participation, and for 2 months following the last dose of study medications (participant can resume oral birth control pills for effective birth control measures after post-treatment biopsy is done). Effective birth control methods during treatment are: copper and Mirena intrauterine device (IUD), diaphragm/cervical cap/shield, spermicide, contraceptive sponge, condoms. Tubal Ligation is an acceptable method of birth control. Women of childbearing potential must have a negative pregnancy test within five days before starting study medications. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.
* Willingness to avoid exposing breast skin to natural or artificial sunlight (i.e. tanning beds) for the duration of the study.
* Participants must have acceptable organ and marrow function as judged by treating physician's evaluation of baseline laboratory data.
* Negative pregnancy (serum or urine) test if of childbearing potential and/or follicle stimulating hormone (FSH) to verify menopausal status.

Exclusion Criteria:

* Clinically suspicious mass/lesions
* Breast cancer in the past 5 years.
* Patients with any history of venous thromboembolic disease, regardless of timeframe (history of varicose veins and superficial phlebitis is allowed).
* Current pregnancy or lactation.
* History of other prior breast cancer-specific therapy within the previous 2 years (chemotherapy, anti-HER2 agents, endocrine agents, everolimus, CDK4-6 inhibitors).
* Cytotoxic chemotherapy for any indication in last 2 years.
* Prior use of selective estrogen receptor modulator (SERMS) or AIs including tamoxifen, raloxifene, anastrozole, letrozole, or exemestane for prevention or therapy within the past 5 years unless:

  * Use was less than 6 months duration in the past 5 years and not used in the 1 year prior to enrollment, or
  * Use was no greater than 2 months duration in the past 1 year and not used in the 6 months prior to enrollment.
* Exogenous sex steroid, including oral contraceptive pill use within 1 month prior to pretreatment breast biopsy. Use of vaginally administered estrogens and hormone coated IUD such as Mirena is permitted.
* History of any prior ipsilateral breast radiotherapy. Previous unilateral radiation of the contralateral side is allowed.
* Skin lesions on the breast that disrupt the stratum corneum (e.g., eczema, ulceration).
* History of endometrial neoplasia
* Current smoker. Cessation for at least 6 weeks
* Current users of potent inhibitors of tamoxifen metabolism. The potent inhibitors of tamoxifen metabolism are: bupropion, cinacalcet, fluoxetine, paroxetine, quinidine.
* Participants may not be receiving any other investigational agents within 90 days of enrollment or during this study.
* History of allergic reactions to tamoxifen.
* Uncontrolled intercurrent illness that in the judgement of the treating physician would make them unsuitable for study participation
* Current use of anticoagulation medications.
* Patients who are breastfeeding.
* Hemoglobin < 10 g/dL (within 30 days of randomization).
* Leukocytes < 3,000/microliter (within 30 days of randomization).
* Platelets < 100,000/microliter (within 30 days of randomization).
* Total bilirubin > 1.5 x institutional upper limit of normal (ULN) (within 30 days of randomization).
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase (SGOT) > 1.5 x ULN (within 30 days of randomization).
* Alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) > 1.5 x ULN (within 30 days of randomization).
* Alkaline phosphatase, S > 1.5 x ULN (within 30 days of randomization).
* Albumin, S > 1.5 x ULN (within 30 days of randomization).
* Protein, total, S > 1.5 x ULN (within 30 days of randomization).
* Creatinine > 1.5 x ULN (within 30 days of randomization).
* Antithrombin III <80% of normal.
* Fibrinogen >1000 mg/dL.
* Patients who are taking any medications, herbal products, or over the counter (OTC) products that are moderate or strong CYP2D6 inhibitors or CYP3A inducers. Patients should also refrain from starting any drug or product with these properties during the study. This is to avoid any potential interactions with tamoxifen or 4-OHT.
* Clinically significant arrhythmia requiring ongoing medication for control / treatment, especially those with high risk of QT prolonging effects.
* Identification of a clinically suspicious mass on examination.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
The purpose of this research is to evaluate short-term changes in background breast tissue induced by oral tamoxifen or 4-OHT gel in women with atypical hyperplasia or lobular carcinoma in situ (LCIS). | 48 months
  Treatment Evaluation/Measurement of Effect

CONTACTS AND LOCATIONS:
Overall Officials: Amy Degnim, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Northwestern University, Evanston, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - MD Anderson Cancer center at Cooper, Camden, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-29): https://cdn.clinicaltrials.gov/large-docs/56/NCT04570956/Prot_SAP_001.pdf
  • Informed Consent Form (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT04570956/ICF_002.pdf